CLINICAL TRIAL: NCT03897088
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Clinical Study to Assess the Efficacy and Safety of Tildrakizumab in the Treatment of Moderate to Severe Plaque Psoriasis of the Scalp
Brief Title: Efficacy and Safety of Tildrakizumab in the Treatment of Scalp Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TILD-18-20
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2022-05

CONDITIONS: Scalp Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tildrakizumab (Experimental)
  Interventions: Drug: PART 1: Double-blind Placebo-controlled; Drug: PART 2: Double-blind Active Treatment Extension
- Placebo (Placebo Comparator)
  Interventions: Drug: PART 1: Double-blind Placebo-controlled
- PART 3: Observational Safety Follow-up (No Intervention): The subjects will not receive study treatment during the follow-up period

INTERVENTIONS:
Drug: PART 1: Double-blind Placebo-controlled — all eligible subjects will receive either tildrakizumab or placebo
  Arms: Placebo; Tildrakizumab
Drug: PART 2: Double-blind Active Treatment Extension — subjects initially on placebo will be switched over to receive tildrakizumab while subjects initially on tildrakizumab will continue to receive tildrakizumab as per defined schedule
  Arms: Tildrakizumab

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of tildrakizumab in the treatment of moderate to severe psoriasis of the scalp.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should be 18 years or older at the time of signing the informed consent during the Screening visit.
2. Subjects with a clinical diagnosis of chronic plaque psoriasis of at least 6 months (as determined by-subject interview and confirmation of diagnosis through physical examination by Investigator).
3. Subjects must have moderate to severe plaque psoriasis of the scalp at Screening and at Baseline, defined by:

   * Scalp Investigator Global Assessment (IGA) of ≥3
   * Psoriasis Scalp Severity Index (PSSI) score of ≥12
   * ≥30% or scalp surface area affected.
4. Subject must have moderate to severe plaque psoriasis at Screening and Baseline defined by

   * Physician Global Assessment for Skin (PGA-S) of at least moderate severity (score of ≥3 on a 5-pointer scale)
   * PASI score of ≥12
   * Body Surface Area (BSA) involvement of >10%
5. Subjects must be considered candidates for systemic therapy, meaning scalp psoriasis inadequately controlled by topical treatments (corticosteroids), and/or phototherapy, and/or previous systemic therapy.
6. Subjects has a negative evaluation for tuberculosis (TB) within 4 weeks before initiating study treatment, defined as a negative QuantiFERON® test. Subjects with a positive or 2 successive indeterminate. QuantiFERON® tests are allowed if they have all of the following:

   * No history of active TB or symptoms of TB.
   * A posterior-anterior chest radiogram (with associated report available at study center) performed within 3 months of Screening with no evidence of active TB (or of any other pulmonary infectious diseases).
   * If prior latent TB infection (LTBI), must have history of adequate prophylaxis (per local standard of care).
   * If presence of LTBI is established, then treatment according to local country guidelines must have been followed for 4 weeks prior to inclusion in the study.

   A maximum of 2 QuantiFERON® tests are allowed. A re-test is only permitted if the first is indeterminate; the result of the second test will then be used.
7. Subjects are unlikely to conceive, as indicated by at least one "Yes" answer to the following questions:

   * Subject is a male.
   * Subject is a female and agrees to abstain from heterosexual activity OR use a highly effective method of contraception as per Appendix 7.
   * Male subjects with female partners of childbearing potential who are not using birth control as described above must use a barrier method of contraception (eg, condom) if not surgically sterile (ie, vasectomy).
   * Subject is a surgically sterilized female or is documented to be postmenopausal. For contraceptive guidance see Appendix 7.
8. For women of childbearing potential, a negative serum pregnancy test at Screening and a negative urine pregnancy test within 24 hours prior to Day 1 and on subsequent visits at which study treatment doses are scheduled.
9. Subjects must have results of a physical examination within normal limits or clinically acceptable limits to the Investigator prior to Day 1. The Investigator is encouraged to consult with the Medical Monitor (or appropriate designee) if there are questions regarding the significance of any out-of-range values.
10. Subjects must be capable of giving signed informed consent as described in Appendix 2, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

1. Subjects who have laboratory abnormalities at Screening including any of the following:

   * Alanine aminotransferase or aspartate aminotransferase ≥2.5 × the upper limit of normal
   * Creatinine ≥2 × the upper limit of normal
   * Serum direct bilirubin ≥1.5 mg/dL
   * White blood cell count <3.0×103/μL
   * Any other laboratory abnormality, which, in the opinion of the Investigator, will prevent the subject from completing the study or will interfere with the interpretation of the study results.
2. Subjects who have predominantly non-plaque forms of psoriasis specifically erythrodermic psoriasis, predominantly pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new-onset guttate psoriasis.
3. Women of childbearing potential who are pregnant, intend to become pregnant (within 6 months of completing the study), or are lactating.
4. Subjects with any infection or history of recurrent infection requiring treatment with systemic antibiotics within 2 weeks prior to Screening, or severe infection (eg, pneumonia, cellulitis, bone or joint infections) requiring hospitalization or treatment with intravenous (IV) antibiotics within 6 weeks prior to Screening.
5. Subjects with any previous use of tildrakizumab or other IL-23/Th-17 pathway inhibitors, including p40, p19 and IL-17 antagonists for psoriasis.

   • Prior use of TNF-alpha inhibitors with a wash-out period of 12 weeks would be allowed. However, the number of subjects with prior use of TNF-alpha inhibitors would be capped at 40% and the analysis will be stratified based on prior use of these biologics.
6. Subjects with a positive human immunodeficiency virus test result, hepatitis B surface antigen, or hepatitis C virus test result.
7. Subjects with a prior malignancy or concurrent malignancy (excluding successfully treated basal cell carcinoma, squamous cell carcinoma of the skin in situ, squamous cell carcinoma of skin with no evidence of recurrence within 5 years or carcinoma in situ of the cervix that has been adequately treated).
8. Subjects who have received live viral or bacterial vaccination within 4-weeks prior to Baseline or who intend to receive live viral or bacterial vaccination during the study.
9. Subjects who are currently participating in another interventional clinical study or has participated in an interventional clinical study within 5-half-lives (of the drug) to wash-out prior to randomization (Subjects participating in observational studies or non-interventional registry studies may be included in the study).
10. Subjects or a family member is among the personnel of the study center or Sponsor/designee staff directly involved with this study.
11. Subjects who have any concomitant medical condition which in the opinion of the Investigator could affect the study outcome or present an unacceptable risk.
12. Subjects who were hospitalized due to an acute cardiovascular event (such as myocardial infarction, cerebrovascular accident, cardiovascular illness [eg, angina pectoris], or cardiovascular surgery [such as coronary artery bypass grafting]) within 6 months before Screening.
13. Subjects who, in the opinion of the Investigator, will not be a reliable participant in the study and those who can confound the results of the study.
14. Subjects who have a history of alcohol or drug abuse in the previous year.
15. Subjects who have high risk of suicidality at the Screening assessment based on Investigator's judgment or, if appropriate, as indicated by a response of "yes" within the last 12 months to Questions 4 or 5 in the suicidal ideation section, or any positive response in the behavioral section of the Columbia-Suicide Severity Rating Scale
16. Subjects with any other clinically significant laboratory abnormality, which, in the opinion of the Investigator, will prevent the subject from completing the study or will interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (19):
  - SPARC Site 18, Encinitas, California
  - SPARC Site 7, Fountain Valley, California
  - SPARC Site 3, Fremont, California
  - SPARC Site 12, Huntington Beach, California
  - SPARC Site 9, Los Angeles, California
  - SPARC Site 2, Los Angeles, California
  - SPARC Site 14, Santa Monica, California
  - SPARC Site 21, Coral Gables, Florida
  - SPARC Site 19, Margate, Florida
  - SPARC Site 5, Sweetwater, Florida
  - SPARC Site 13, East Windsor, New Jersey
  - SPARC Site 4, Forest Hills, New York
  - SPARC Site 16, New York, New York
  - SPARC Site 01, Beachwood, Ohio
  - SPARC Site 20, Portland, Oregon
  - SPARC Site 8, Johnston, Rhode Island
  - SPARC Site 17, Cypress, Texas
  - SPARC Site 11, Houston, Texas
  - SPARC Site 6, Webster, Texas
- Australia (6):
  - SPARC Site 23, Kogarah, New South Wales
  - SPARC Site 27, Kogarah, New South Wales
  - SPARC Site 26, Woolloongabba, Queensland
  - SPARC Site 25, Carlton, Victoria
  - SPARC Site 24, East Melbourne, Victoria
  - SPARC Site 22, Fremantle, Western Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: All eligible subjects will receive Placebo injections upto week 4. At Week 16, all the subjects from this arm were switched to receive Tildrakizumab upto week 52.
- Tildrakizumab: All eligible subjects will receive Tildrakizumab upto week 52.
Period: Overall Study
Arm/Group | Placebo | Tildrakizumab
Started | 114 | 117
Completed | 88 | 86
Not Completed | 26 | 31
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Lost to Follow-up | 7 | 15
Not completed — Sponsor Decision | 1 | 2
Not completed — COVID-19 | 2 | 0
Not completed — Other | 3 | 0
Not completed — Non-compliance with Study Drug | 1 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: All eligible subjects will receive Placebo injections upto week 4. At Week 16, all the subjects from this arm were switched to receive Tildrakizumab upto 52.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tildrakizumab | Total
Number analyzed (Participants) | 114 | 117 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (12.96) | 45.6 (15.27) | 45.2 (14.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 46 | 97
  Male | 63 | 71 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 42 | 87
  Not Hispanic or Latino | 69 | 75 | 144
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects With Investigator Global Assessment Mod 2011 (Scalp) Score of "Clear" and "Almost Clear" With at Least 2-point Reduction From Baseline at Week 16
Time Frame: Week 16
Measure: Number; unit: proportion of subjects
Groups:
- Placebo Comparator: Placebo: Subjects will receive Placebo injections upto week 4. At Week 16, all the subjects from this arm were switched to receive Tildrakizumab upto week 52.
- Tildrakizumab: Subjects will receive Tildrakizumab upto week 52
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 82 | 89
proportion of subjects | 0.073 | 0.494
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Week 16; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel

2. Primary Outcome: The Percentage of Subjects With Incidence, Seriousness and Severity of All Adverse Events.
Time Frame: Week 72
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Percentage of participants
  Incidence of TEAEs | 51.8 | 53
  Serious TEAEs | 3.5 | 2.6
  Severity - Mild | 45.6 | 40.1
  Severity - Moderate | 21.1 | 18.8
  Severity- Severe | 1.7 | 0.8

3. Primary Outcome: The Percentage of Subjects With Severe Infections, Whether or Not Reported as a Serious Event
Description: defined as any infection meeting regulatory definition of serious adverse event, or any infection requiring intravenous antibiotics whether or not reported as a serious event as per the regulatory definition.
Time Frame: Week 72
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Percentage of participants | 0 | 0

4. Primary Outcome: The Percentage of Subjects With Malignancies (Excluding Carcinoma in Situ of the Cervix).
Time Frame: Week 72
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Percentage of participants | 0 | 1.71

5. Primary Outcome: The Percentage of Subjects With Melanoma Skin Cancer.
Time Frame: Week 72
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Percentage of participants | 0 | 0

6. Primary Outcome: The Percentage of Subjects With Major Adverse Cardiovascular Events
Time Frame: Week 72
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Percentage of participants | 1.75 | 0.85

7. Primary Outcome: The Percentage of Subjects With Study Treatment-related Hypersensitivity Reactions (eg, Anaphylaxis, Urticaria, Angioedema, Etc.).
Time Frame: Week 72
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Percentage of participants | 1.75 | 0.85

8. Primary Outcome: The Percentage of Subjects With Injection Site Reactions (eg, Pain, Erythema, Edema Etc).
Time Frame: Week 72
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Percentage of participants | 0.88 | 0

9. Primary Outcome: The Percentage of Subjects With Non-melanoma Skin Cancer
Time Frame: Week 72
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Percentage of participants | 0 | 2

10. Secondary Outcome: The Proportion of Subjects With at Least 90% Improvement From Baseline in the Psoriasis Scalp Severity Index at Week 16
Time Frame: Week 16
Measure: Number; unit: proportion of subjects
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
proportion of subjects | 0.044 | 0.56
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Week 16; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel

11. Secondary Outcome: Mean Percentage Change in Psoriasis Scalp Severity Index Score From Baseline to Week 16.
Description: Psoriasis Scalp Severity Index (PSSI) use a 5-point scale to grade the 3 clinical parameters (erythema, thickness, and scaling) in the same way as the Psoriasis Area Severity Index (PASI), but for scalp only. The parameter scores are summed and multiplied by an integer (0-6) that represents the area of affected scalp. The score ranges from 0-72. Outcome measures percentage change in score from baseline. Lesser the score, better is the outcome.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: Mean percent change
Groups:
- Placebo Comparator: Placebo: Subjects will receive Placebo injections upto week 4. At Week 16, all the subjects from this arm were switched to receive Tildrakizumab upto week 52
  .
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 107 | 110
Mean percent change | -21.84 (35.577) | -79.81 (30.434)
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Week 16; Test type: Superiority; p < 0.00001, Mixed Models Analysis

12. Secondary Outcome: The Proportion of Subjects Achieving Psoriasis Scalp Severity Index 75 at Week 16
Description: Psoriasis Area and Severity Index is use a 5-point scale to grade the 3 clinical parameters (erythema, thickness, and scaling). The PASI includes scores on erythema, thickness, scaling, and percentage of body surface area (BSA) affected. The parameter scores are summed and multiplied by an integer (0-6) that represents the area of affected scalp. The score ranges from 0-72. Outcome measures percentage change in score from baseline. Current outcome measures proportion of subjects achieving 75% improvement from baseline.
Time Frame: Week 16
Measure: Number; unit: proportion of subjects
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
proportion of subjects | 0.105 | 0.709
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Week 16; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel

13. Secondary Outcome: The Proportion of Subjects Achieving Psoriasis Scalp Severity Index 100 at Week 16
Description: Psoriasis Scalp Severity Index (PSSI) use a 5-point scale to grade the 3 clinical parameters (erythema, thickness, and scaling) in the same way as the Psoriasis Area Severity Index (PASI), but for scalp only. The parameter scores are summed and multiplied by an integer (0-6) that represents the area of affected scalp. The score ranges from 0-72. Outcome measures percentage change in score from baseline. Lesser the score, better is the outcome. Current outcome measures 100% improvement in PSSI from baseline.
Time Frame: Week 16
Measure: Number; unit: proportion of subjects
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
proportion of subjects | 0.026 | 0.376
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Week 16; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel

14. Secondary Outcome: Mean Percentage Change in Scalp Surface Area (SSA) Involvement From Baseline to Week 16
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: Mean percent change in SSA
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 107 | 110
Mean percent change in SSA | -15.20 (31.473) | -76.39 (35.179)
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Week 16; Test type: Superiority; p < 0.00001, Mixed Models Analysis

15. Secondary Outcome: Time to 75% Reduction in Psoriasis Scalp Severity Index During 16-week Placebo-controlled Treatment Period.
Description: Psoriasis Scalp Severity Index (PSSI) use a 5-point scale to grade the 3 clinical parameters (erythema, thickness, and scaling) in the same way as the Psoriasis Area Severity Index (PASI), but for scalp only. The parameter scores are summed and multiplied by an integer (0-6) that represents the area of affected scalp. The score ranges from 0-72. Outcome measures percentage change in score from baseline.
  Current outcome measure is time to PSSI 75. Lesser the time required, better is the effect of drug.
Time Frame: Week 16
Measure: Median (Inter-Quartile Range); unit: Time (days)
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Time (days) | NA [NA to NA] — Not estimable due to insufficient number of non-censored observations | 59 [54 to 113]
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Test type: Superiority; p < 0.00001, Kaplan-Meier Estimates — Log Rank Test p-Value

16. Secondary Outcome: Time to Investigator Global Assessment Mod 2011 (Scalp ) Response During the 16-week Placebo-controlled Treatment Period.
Description: Investigator Global Assessment Mod 2011 (Scalp) is a 5-point scale that is static (refers exclusively to the subject's disease state at the time of the assessments, and does not attempt a comparison with any of the subject's previous disease states, whether at baseline or at a previous visit). Score ranges from 0-4. lower the score is better. Traetment success is considered when IGA Mod 2011 (Scale) is 0 or 1 with 2 point reduction from baseline score. current outcome measures time to treatment success.
Time Frame: Week 16
Measure: Median (Inter-Quartile Range); unit: Time (days)
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 82 | 89
Time (days) | NA [NA to NA] — Not estimable due to insufficient number of non-censored observations | 86 [57 to 115]
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Test type: Superiority; p < 0.00001, Kaplan-Meier Estimates — Log Rank Test p-Value

17. Secondary Outcome: Proportion of Subjects Achieving a 4-point Reduction in Itch Numeric Rating Scale Score From Baseline to Week 16
Time Frame: Week 16
Measure: Number; unit: Proportion of subjects
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 102 | 101
Proportion of subjects | 0.147 | 0.545
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel

18. Secondary Outcome: The Proportion of Subjects Achieving Psoriasis Area and Severity Index (PASI) 75, Psoriasis Area and Severity Index 90, and Psoriasis Area and Severity Index 100 at Week 16
Description: Psoriasis Area and Severity Index is use a 5-point scale to grade the 3 clinical parameters (erythema, thickness, and scaling). The PASI includes scores on erythema, thickness, scaling, and percentage of body surface area (BSA) affected. The parameter scores are summed and multiplied by an integer (0-6) that represents the area of affected scalp. The score ranges from 0-72. Outcome measures percentage change in score from baseline. Current outcome measures proportion of subjects achieving 75%, 90% and 100% improvement from baseline, respectively.
Time Frame: Week 16
Measure: Number; unit: Proportion of subjects
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Proportion of subjects
  PASI-75 | 0.079 | 0.667
  PASI-90 | 0.026 | 0.41
  PASI-100 | 0.009 | 0.162
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; PASI-75; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; PASI-90; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; PASI-100; Test type: Superiority; p = 0.00004, Cochran-Mantel-Haenszel

19. Secondary Outcome: The Proportion of Subjects With Physician's Global Assessment Score (Whole Body) Score of "Clear" or "Almost Clear" With at Least a 2-point Reduction From Baseline to Week 16
Time Frame: Week 16
Measure: Number; unit: Proportion of subjects
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Proportion of subjects | 0.062 | 0.556
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Week 16; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel

20. Secondary Outcome: Mean Percentage Change in Total Body Surface Area (BSA) Involvement From Baseline to Week 16
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: Mean percent change in BSA
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 107 | 110
Mean percent change in BSA | 0.19 (39.039) | -70.17 (33.443)
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Week 16; Test type: Superiority; p < 0.00001, Mixed Models Analysis

21. Secondary Outcome: The Proportion of Subjects With Investigator Global Assessment (Scalp Only) Score of "Clear" and "Almost Clear" With at Least 2-point Reduction From Baseline at Week 16.
Time Frame: Week 16
Measure: Number; unit: Proportion of subjects
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Proportion of subjects | 0.106 | 0.684
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Week 16; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel

22. Secondary Outcome: The Proportion of Subjects With Investigator Global Assessment Mod 2011 Score (Whole Body) of "Clear" and "Almost Clear" With at Least 2-point Reduction From Baseline at Week 16
Time Frame: Week 16
Measure: Number; unit: Proportion of subjects
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 82 | 89
Proportion of subjects | 0.038 | 0.545
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel — Week 16

23. Secondary Outcome: The Proportion of Subjects With IGA Mod 2011 (Scalp) Score of "Clear" and "Almost Clear" With at Least 2-point Reduction From Baseline
Time Frame: Week 12
Measure: Number; unit: Proportion of subjects
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 82 | 89
Proportion of subjects | 0.049 | 0.461
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Week 12; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel

24. Secondary Outcome: The Proportion of Subjects With at Least 90% Improvement From Baseline in the Psoriasis Scalp Severity Index
Time Frame: week 12
Measure: Number; unit: Proportion of subjects
Arm/Group | Placebo Comparator: Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
Proportion of subjects | 0.018 | 0.427
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Tildrakizumab; Week 12; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel

25. Secondary Outcome: Change in Investigator Global Assessment Mod 2011 (Scalp) From Baseline at Week 52
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Subjects will receive Placebo injections upto week 4. At Week 16, all the subjects from this arm were switched to receive Tildrakizumab upto week 52.
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 68 | 77
Participants
  1 = Worsen by 1 | 0 | 0
  0 = No Change | 1 | 2
  -1 = Improve by 1 | 14 | 13
  -2 = Improve by 2 | 9 | 9
  -3 = Improve by 3 | 38 | 48
  -4 = Improve by 4 | 6 | 5

26. Secondary Outcome: Change in IGA Mod 2011 (Whole-body) From Baseline at Week 52
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 65 | 76
Participants
  1 = Worsen by 1 | 0 | 0
  0 = No Change | 6 | 5
  -1 = Improve by 1 | 15 | 18
  -2 = Improve by 2 | 15 | 18
  -3 = Improve by 3 | 26 | 33
  -4 = Improve by 4 | 3 | 2

27. Secondary Outcome: Mean Change in Psoriasis Scalp Severity Index Score From Baseline at Week 52
Description: as for outcome 11
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
score on a scale | -30.4 (15.39) | -31.1 (13.96)

28. Secondary Outcome: Change From Baseline in Investigator Global Assessment (Scalp Only) at Week 52
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 97 | 100
Participants
  1 = Worsen by 1 | 1 | 0
  0 = No Change | 4 | 3
  -1 = Improve by 1 | 8 | 8
  -2 = Improve by 2 | 18 | 14
  -3 = Improve by 3 | 58 | 66
  -4 = Improve by 4 | 8 | 9

29. Secondary Outcome: Change From Baseline in Scalp Itch Numeric Rating Scale (NRS) Score at Week 52
Description: The Scalp Itch NRS is a self-administered, single item questionnaire with response options from 0=No Itch to 10=Worst itch imaginable. A higher score on the NRS corresponds to greater scalp itch severity.
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
score on a scale | -5.0 (3.04) | -4.7 (3.04)

30. Secondary Outcome: Mean Change in PASI Score From Baseline at Week 52
Description: Psoriasis Area Severity Index (PASI) use a 5-point scale to grade the 3 clinical parameters (erythema, thickness, and scaling). The parameter scores are summed and multiplied by an integer (0-6) that represents the area of affected scalp. The score ranges from 0-72. Outcome measures percentage change in score from baseline. Lesser the score, better is the outcome.
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
score on a scale | -16.43 (7.901) | -16.84 (6.072)

31. Secondary Outcome: Change in Physician Global Assessment for Skin (Whole Body) From Baseline at Week 52
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 96 | 100
Participants
  1 = Worsen by 1 | 1 | 6
  0 = No Change | 8 | 12
  -1 = Improve by 1 | 15 | 12
  -2 = Improve by 2 | 26 | 27
  -3 = Improve by 3 | 38 | 49
  -4 = Improve by 4 | 8 | 6

32. Other Pre Specified Outcome: Change From Baseline in Dermatology Life Quality Index Score (Total and 6 Domain Scores) at Measured Time Points Through Week 52
Description: The DLQI questionnaire is used to assess treatment response on the subject's quality of life. The aim of this questionnaire is to measure how much the skin condition has affected the subject's life during the previous week.
  Subjects are asked to recall their experiences during the previous week by responding to 10 questions. The questionnaire is self-explanatory and handed to the subject who is asked to fill it in without the need for a detailed explanation. DLQI is calcualted by summing the score of each question resulting in a maximum of 30 and minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Tildrakizumab
Number analyzed (Participants) | 114 | 117
score on a scale
  Total | -12.5 (6.74) | -11.5 (7.51)
  Symptoms and Feelings | -3.4 (1.27) | -3.2 (1.61)
  Daily Activities | -2.8 (1.62) | -2.6 (1.90)
  Leisure | -2.4 (1.93) | -2.2 (2.03)
  Work and School | -0.9 (1.09) | -0.9 (1.17)
  Personal Relationships | -1.8 (1.86) | -1.7 (1.97)
  Treatment | -1.1 (1.26) | -0.9 (1.12)

ADVERSE EVENTS:
Time Frame: 72 weeks
Groups:
- Placebo: Subjects will receive Placebo injections upto week 4.
- Placebo to Tildrakizumab: At week 16, subjects initially randomized to placebo were switched to receive Tildrakizumab upto Week 52
Arm/Group | Placebo | Placebo to Tildrakizumab | Tildrakizumab
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/114 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/114 | 4/114 | 3/117
Other Adverse Events (participants affected / at risk) | 13/114 | 17/114 | 46/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=114) | Placebo to Tildrakizumab (N=114) | Tildrakizumab (N=117)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=114) | Placebo to Tildrakizumab (N=114) | Tildrakizumab (N=117)
Nasopharyngitis (Infections and infestations) | 1 | 5 | 5
Covid-19 (Infections and infestations) | 0 | 4 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 3
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 3
Influenza (Infections and infestations) | 0 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 2
Sars-Cov-2 Test Positive (Investigations) | 0 | 2 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1
Blood Triglycerides Increased (Investigations) | 2 | 0 | 0
Weight Increased (Investigations) | 0 | 0 | 2
Headache (Nervous system disorders) | 4 | 2 | 3
Sciatica (Nervous system disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 2 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 2
Seasonal Allergy (Immune system disorders) | 1 | 0 | 2
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 3
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03897088/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03897088/SAP_001.pdf